CLINICAL TRIAL: NCT06135493
Title: Efficacy of Losartan in the Prevention of Paclitaxel-induced Peripheral Neuropathy in Breast Cancer Patients.
Brief Title: Prevention of Paclitaxel-induced Peripheral Neuropathy in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Alaa Mahmoud Ahmed Shawqy Mahmoud, Principle Invistigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC-FPFUE-30/2023
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Neuropathy Due to Chemotherapy
Keywords: Paclitaxel; Breast Cancer; Peripheral Neuropathy
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases | interventions — Losartan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): These patients will receive standard-of-care management for chemotherapy-induced nausea and vomiting
- Intervention arm (Experimental): These patients will receive standard-of-care management for chemotherapy-induced nausea and vomiting plus losartan 100mg
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — Using losartan to prevent paclitaxel-induced peripheral neuropathy
  Arms: Intervention arm

SUMMARY:
Paclitaxel-induced peripheral neuropathy (PIPN) is one of the most dose-limiting side effects; it causes patients discomfort and pain and sometimes causes the termination of the chemotherapy cycles, leading to treatment failure. A lot of interventions have been tried to prevent PIPN, ensure complete administration of the chemotherapy cycles, and increase the survival rate. One of the promising interventions in the prevention of PIPN is Losartan. Losartan is an angiotensin receptor blocker (ARBs) and is used to treat hypertensive patients. There is strong evidence from different preclinical studies and retrospective cohort studies that Losartan has a neuroprotective effect.

The purpose of our study is to investigate the efficacy of Losartan in the prevention of peripheral neuropathy associated with Paclitaxel treatment in Breast Cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Females older than 18 years diagnosed with biopsy-confirmed breast cancer (Early breast cancer eligible for adjuvant or neoadjuvant) who are scheduled to receive paclitaxel 80 mg/m2.

Exclusion Criteria:

* Known hypersensitivity to Losartan.
* Not Known Hypertensive patients
* Not Known Diabetic patients
* Treatment with Losartan/ARBs/ACE-I prior to the study.
* Previous neuropathy
* Renal impairment (Serum creatinine > 2 mg/dl)
* Significant liver disease: liver enzymes 2 folds the upper normal limit
* Metastatic breast cancer
* Pregnancy or lactation
* Taking other medication for neuropathic pain
* Significant Hypotension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Development of paclitaxel-induced peripheral neuropathy | 12 weeks
  Incidence and grading of paclitaxel-induced peripheral neuropathy (PIPN)

SECONDARY OUTCOMES:
Patient QOL | 12 weeks
  Patient quality of life will be assessed by Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT/GOG-NTX)
Pain Severity | 12 Weeks
  Pain intensity will be assessed through Visaul Analogue Scale Scale 0-10
Serum biomarker | 12 weeks
  Level of Nerve growth factor (NGF) in Serum

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Cancer Comprehensive Center of the National Cancer Institute, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No